CLINICAL TRIAL: NCT06955520
Title: Vonaprazan Versus Esomeprazole for Healing of LA Grade B or Higher Esophagitis After POEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFCNet 1
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded for this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- To assess the efficacy of vonapraprazon 20mg better than esomeprazole drug (Active Comparator): healing rate will be checked during endoscopy at 8 weeks
  Interventions: Drug: Vonoprazan
- To see the healing rate of grade B esophagitis (Placebo Comparator): healing rate will be checked during endoscopy at 8 weeks in patients receiving esomeprazole 40mg
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: Vonoprazan — a potassium-competitive acid blocker (P-CAB), offers superior acid suppression and may provide enhanced healing in post-POEM reflux esophagitis.
  Other Names: per oral endoscopy myotomy
  Arms: To assess the efficacy of vonapraprazon 20mg better than esomeprazole drug
Drug: Esomeprazole 40mg — It is a proton pump inhibitor which reduces the excessive acid secretion in the stomach and it heals grade B esophagitis (>5mm ulcer between two mucosal folds in esophagus)
  Other Names: per oral endoscopy myotomy
  Arms: To see the healing rate of grade B esophagitis

SUMMARY:
Peroral Endoscopic Myotomy (POEM) is a well-established treatment for achalasia; however, it is frequently associated with gastroesophageal reflux disease (GERD), with many patients developing LA grade B or higher esophagitis. Proton pump inhibitors (PPIs) like Esomeprazole are the standard treatment, but Vonaprazan, a potassium-competitive acid blocker (P-CAB), offers superior acid suppression and may provide enhanced healing in post-POEM reflux esophagitis.

Primary Objective:

• To compare the healing rates of LA grade B or higher reflux esophagitis at 8 weeks in patients receiving Vonaprazan 20 mg versus Esomeprazole 40 mg.

Secondary Objectives

* To assess improvement in reflux symptoms using the GERD-Q score at 8 weeks.
* To evaluate the incidence of adverse events in each treatment group.

DETAILED DESCRIPTION:
Study Type:

• Randomized, Open-Label, Two-Arm, Non-Inferiority Trial

Randomization and Blinding:

* Randomization: 1:1 ratio between Vonaprazan 20 mg and Esomeprazole 40 mg.
* Stratification: Based on LA grade (B vs. C/D) at baseline.
* Blinding: Open-label study, but outcome assessors will be blinded.

Study Timeline:

1. All post-POEM patients receive Esomeprazole 40 mg for 2 months.
2. PPI is discontinued for 1 month (to allow reflux esophagitis to develop if persistent GERD exists).
3. At 3 months post-POEM, patients with LA grade B or higher esophagitis (on follow-up endoscopy) are randomized to either Vonaprazan 20 mg or Esomeprazole 40 mg for 8 weeks.
4. At 8 weeks post-randomization (5 months post-POEM), healing of esophagitis is assessed.

Study Arms:

* Arm A: Vonaprazan 20 mg once daily for 8 weeks
* Arm B: Esomeprazole 40 mg once daily for 8 weeks

Study Procedures:

Baseline Assessment (3 Months Post-POEM, Before Randomization)

* Upper GI Endoscopy: Confirmation of LA grade B or higher reflux esophagitis.
* GERD-Q Score assessment.
* Randomization to Vonaprazan 20 mg or Esomeprazole 40 mg. Follow-Up (Week 4 - Interim Visit)
* GERD-Q Score assessment.

End-of-Treatment (Week 8 - Final Visit, 5 Months Post-POEM)

* Upper GI Endoscopy to assess healing of reflux esophagitis.
* GERD-Q Score reassessment.
* Final adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of POEM for achalasia
* Endoscopic confirmation of LA grade B, C, or D reflux esophagitis at 3 months post-POEM
* GERD symptoms (heartburn, regurgitation) for ≥4 weeks
* Willingness to provide informed consent and comply with study procedures

Exclusion Criteria:

* History of prior anti-reflux surgery
* Presence of Barrett's esophagus, esophageal stricture, or malignancy
* Severe gastroparesis or esophageal motility disorder unrelated to achalasia
* Pregnancy or breastfeeding
* Severe hepatic or renal impairment (ALT/AST >3× ULN, eGFR <30 mL/min)
* Regular use of NSAIDs, steroids, or anticoagulants affecting esophageal healing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
• Endoscopic healing of reflux esophagitis at 8 weeks (absence of LA grade B or higher esophagitis). | 8 weeks
  This can be find during endoscopy test

SECONDARY OUTCOMES:
• Improvement in GERD-Q scores at 8 weeks | 8 weeks
  GERD questionnaire can be calculated based on heart burn , regurgitation symptom scores which is scaled like 1 is very low symptoms, 5 is worse symptoms (outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MD DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No